CLINICAL TRIAL: NCT02824601
Title: Does Supplemental Photodynamic Therapy Optimize the Disinfection of Bacteria and Endotoxins in One-visit and Two-visit Root Canal Therapy? A Randomized Clinical Trial
Brief Title: Photodynamic Therapy in Endodontic Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Frederico Canato Martinho, DDS, Ms, PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 43555515.9.0000.0077
Record Dates: First submitted 2016-06-24; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Endodontic Disease
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Lasers; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- One-visit treatment PDT (Experimental): Intervention: Chemo-mechanical preparation (CMP) was performed by using the single-file reciprocating technique + 2.5% NaOCL and a final rinse with 17% EDTA. Next, the root canals were irrigated with 10 mL of saline solution, with calcium hydroxide medication being neutralized with 0.5% citric acid. Afterwards, the photosensitizer agent (methylene blue 10 mg/mL) was applied to root canals for 60 seconds and submitted to laser with a potency of 60 mW and energy density of 129 J/cm2 for 120 seconds after CMP in the one-visit treatment
  Interventions: Device: Laser
- Two-visit treatment PDT (Experimental): Intervention: Chemo-mechanical preparation (CMP) was performed by using the single-file reciprocating technique + 2.5% NaOCL and a final rinse with 17% EDTA. In the following, 14-day inter-appointment medication with Ca(OH)2 + SSL was placed in the root canal. After 14 days with intracanal medication, the tooth was isolated for surgery and disinfection, including removal of provisional restoration. Next, the root canals were irrigated with 10 mL of saline solution, with calcium hydroxide medication being neutralized with 0.5% citric acid. Afterwards, the photosensitizer agent (methylene blue 10 mg/mL) was applied to root canals for 60 seconds and submitted to laser with a potency of 60 mW and energy density of 129 J/cm2 for 120 seconds after CMP in the one-visit treatment
  Interventions: Device: Laser; Drug: Calcium hydroxide

INTERVENTIONS:
Device: Laser — 1-visit-treatment (n=12): Chemomechanical preparation (CMP) - CMP was performed by using the single-file reciprocating technique + 2.5% NaOCL and 17% EDTA. Methylene blue was applied to root canals for 60 seconds and submitted to laser with a potency of 60 mW and energy density of 129 J/cm2 for 120 seconds after CMP
  Other Names: PDT
Drug: Calcium hydroxide — 2-visit-treatment (n=12): Chemomechanical preparation (CMP) + Ca(OH)2 + SSL medication for 14-days + PDT. CMP was performed by using the single-file reciprocating technique + 2.5% NaOCL and 17% EDTA. Methylene blue was applied to root canals for 60 seconds and submitted to laser with a potency of 60 mW and energy density of 129 J/cm2 for 120 seconds after 14-days of intracanal medication
  Arms: Two-visit treatment PDT

SUMMARY:
This randomized clinical trial evaluated the effectiveness of supplemental photodynamic therapy (PDT) in optimizing the removal of bacteria and endotoxins from primarily infected root canals after one-visit and two-visit treatments.Twenty-four primarily infected root canals with apical periodontitis were selected and randomly divided into one-visit (n=12) and two-visit treatments (n=12). Chemo-mechanical preparation (CMP) was performed by using the single-file reciprocating technique + 2.5% NaOCL and a final rinse with 17% Ethylenediamine tetraacetic acid (EDTA). The photosensitizer agent (methylene blue 10 mg/mL) was applied to root canals for 60 seconds and submitted to laser with a potency of 60 milliwatts (mW) and energy density of 129 J/cm2 for 120 seconds after CMP in the one-visit treatment and after 14-day inter-appointment medication with Ca(OH)2 + saline solution (SSL) in the two-visit treatment. Samples were collected before and after root canal procedures. Endotoxins were quantified by chromogenic limulus amebocyte lysate assay. Culture techniques were used to determine bacterial colony-forming unit counts.

ELIGIBILITY:
Inclusion Criteria:

* single-rooted maxillary ones with primary endodontic infection and showing presence of one root canal and absence of periodontal pockets deeper than 4 mm.

Exclusion Criteria:

* Those who had received antibiotic treatment during the past three months were excluded.
* The teeth that could not be isolated with rubber dam were also excluded.
* Presence of root canal calcification.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in the Determination of Total Cultivable Bacterial Count | At Baseline and after 14-day intracanal medication
  Briefly, the transport media containing the root canal samples were thoroughly shaken for 60 seconds. Serial 10-fold dilutions were made up to 10-4 in tubes containing fastidious anaerobe broth (FAB; Lab M, Bury, UK). Fifty microliters of the serial dilutions was plated onto 5% defibrinated sheep blood fastidious anaerobe agar (FAA; LabM) by using sterile plastic spreaders to culture non-selectively obligate anaerobes and facultative anaerobes. The plates were incubated at 37°C in anaerobic atmosphere for up to 14 days. After this period, colony-forming units (CFUs) were visually quantified for each plate.

SECONDARY OUTCOMES:
Change in the Quantification of Endotoxin Concentration | At Baseline and after 14-day intracanal medication
  The kinetic chromogenic limulus amebocyte lysate (LAL) assay was used for quantification of endotoxins, with Escherichia coli endotoxin being used as standard. For the test, 100 mL of apyrogenic water (reaction blank), five standard endotoxin solutions [0.005-50 endotoxin units (EU/mL)], root canal samples, and positive controls (root canal samples contaminated with a known concentration of endotoxin, i.e. 10 EU/mL) were added to a 96-well apyrogenic plate. The tests were carried out in quadruplicate. The plate was incubated at 37°C±1°C for 10 minutes in a Kinetic reader, which was coupled to a microcomputer by means of a software. Next, 100 mL of chromogenic reagent was added to each well. The software continuously monitored absorbance at 405 nm in each microplate well and automatically calculated the log/log linear correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Frederico C Martinho, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Paulista Júlio de Mesquita Filho, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes